CLINICAL TRIAL: NCT00346138
Title: Deep Lamellar Endothelial Keratoplasty as Surgical Treatment for Corneal Endothelial Decompensation
Brief Title: A Comparison Between Full Thickness and Partial Thickness Corneal Transplantation for Corneal Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000-03
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Fuchs Dystrophy; Corneal Edema
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Edema | interventions — Corneal Transplantation

INTERVENTIONS:
Procedure: Corneal transplantation

SUMMARY:
The objectives of this study are to compare the visual and refractive outcomes of deep lamellar endothelial keratoplasty (DLEK) with penetrating keratoplasty as treatment for certain cases of corneal edema due to endothelial decompensation. Additionally, data will be collected to compare corneal shape, corneal thickness, endothelial cell density, keratocyte density, corneal sensitivity, light scatter, and subjective visual function between the two procedures.

DETAILED DESCRIPTION:
This will be a randomized prospective study. We will enroll patients using the following inclusion and exclusion criteria, based upon the surgeon?s initial complete ophthalmic examination, which includes refraction, keratometry, slit lamp examination, intraocular pressure and corneal thickness measurement, and dilated fundus examination.

Inclusion criteria:

1) Both males and females are eligible 2) Patient age 21 years or older 3) Corneal edema due to endothelial dysfunction 4) Aphakia, pseudophakia, or cataract requiring extraction 5) Visual acuity as measured in standardized fashion (ETDRS chart and appropriate illumination)

1. Study eye; best spectacle-corrected entrance acuity 20/40 or worse
2. Contralateral eye; best spectacle-corrected entrance acuity equal to or better than the study eye and 20/200 or better.

   Exclusion criteria:

   1) Central stromal corneal scars 2) Presence of a filtering bleb 3) History of Herpes simplex or Herpes zoster keratitis 4) Uncontrolled glaucoma 5) Pregnancy. Serum pregnancy testing will be performed within 7 days prior to surgery for women of child-bearing potential

   In the 2-year period, January 2001 to January 2003, 67 PK?s were performed at Mayo Clinic for endothelial dysfunction (e.g., Fuch?s dystrophy or pseudophakic corneal edema) in patients who met the entry criteria for this protocol. During the 2-year enrollment period of this study, we anticipate that up to 50 patients will be enrolled. Appropriate counseling will be done, including a discussion of the potential benefits and risks of the procedures. IRB-approved consent forms will be signed. Enrolled patients will return on a different day (often the day before surgery or the morning of surgery to be performed in the afternoon) for the preoperative Keratogram. Randomization and assignment of the patient to DLEK or PK will occur after the preoperative Keratogram and after the surgeon has accepted a donor cornea from the eye bank for the procedure.

   Keratogram

   The Keratogram consists of a series of tests administered both pre- and post-operatively by trained research personnel who are masked to the patients? particular randomizations. Keratograms will be performed preoperatively and at 1 month (3-6 weeks), 3 months (2-4 months), 6 months (5-7 months), and 1, 2, and 3 years (3 months) postoperatively. The following measurement procedures, to be conducted only on the operated eye, are included in each Keratogram. The equipment to be used is included in parentheses:

   1. Contrast sensitivity with best refraction (Ginsburg contrast sensitivity tester) 2. Straylight meter measurement (Van den Berg straylight meter) 3. Corneal topography map (TMS-2) 4. Corneal profile (Orbscan) 5. Noncontact endothelial photography (Konan Robo) 6. Scatterometry (Mayo scatterometer) 7. Corneal esthesiometry (Belmonte esthesiometer) 8. Confocal microscopy (Tandem Scanning or Confoscan 3 confocal microscope) 9. Quality of visual function questionnaire (NEI-VFQ). This will not be done at the 1week, one month, or 3 month visit.

   Eligibility of Fellow Eyes Fellow eyes in bilateral cases will be eligible to enter the study 4 months or more after the first procedure if these eyes now meet the eligibility criteria (i.e., if the fellow eye now has worse vision than the operated study eye). These eyes will be randomized separately and follow the same protocol, with the exception that the patient may override the randomization if he or she prefers to have one or the other of the 2 procedures. For data analysis, fellow eyes will be considered a separate group.

   Adverse Occurrences For DLEK, adverse occurrences at the time of surgery (such as premature entry into the anterior chamber during recipient lamellar dissection) will require conversion to a standard PK and the patient will be exited from the study. Adverse postoperative occurrences in either surgical group (such as a dislocated disc, uncontrolled rejection, primary graft failure, infection or other adverse events) will be managed by the surgeon according to standard practices. These patients will remain in the study and will have identical follow-up.

   SURGICAL METHODS
   1. DLEK

   Anesthesia:

   Anesthesia options will include monitored, attended, local anesthesia or general orotracheal anesthesia, depending on the particular patient?s desire and comorbid conditions. For local anesthesia a standard retrobulbar and facial nerve block as done for standard PK will be utilized.

   Preparation of recipient:
   1. In the preoperative area, pilocarpine 1%, one drop to operated eye is instilled every five minutes for 3 doses in order to constrict the pupil.
   2. After anesthesia is attained and the eye is prepared and draped, the lid speculum and operating microscope with video recording of each case is brought into position.
   3. Rectus bridle sutures for positioning of the globe are placed as necessary.
   4. A limbal peritomy is performed and the conjunctiva is recessed from the 9:30 to 2:30 o'clock superior limbus.
   5. A limbal incision of the sclera, 1.0 mm peripheral to the limbus and parallel to the limbus, is made with a guarded diamond knife set to 0.35 mm depth. The length of the incision is 9.0 mm or 4.5mm, measured with calipers.
   6. Deep lamellar dissection of the cornea utilizing a crescent blade is performed followed by a stromal dissector spatula.
   7. Paracentesis and Healon injection to maintain the anterior chamber.
   8. Placement of intra-lamellar trephine with trephination of the recipient posterior stromal disc. If a 4.5mm incision was made, then the trephine is used to make an indentation on the corneal surface and the posterior lamellar disc is cut with scissors.
   9. Entry into anterior chamber with a diamond blade at 12 o'clock in the trephination.
   10. Excision of recipient posterior stromal disc and endothelium with corneal scissors and removal of disc from the eye.
   11. Caliper measurement of the diameter of the excised tissue is recorded.
   12. Wound closure and standard phacoemulsification and IOL implantation through a separate incision in patients requiring cataract removal.
   13. Healon is evacuated completely from the anterior chamber with an I/A unit. (eg: Simcoe Needle).
   14. The cornea is covered with a moistened gauze disc.

   Preparation of donor tissue
   1. Donor corneo-scleral tissue is removed from the storage media, endothelium is coated with healon, and the tissue is secured in the Moria artificial anterior chamber.
   2. A deep lamellar dissection pocket is formed in the donor with a crescent blade followed by a stromal dissector spatula.
   3. The donor tissue is placed (endothelial side up) onto the trephination block and the same size trephine (same size as recipient disc tissue diameter) is used to trephine the donor disc.
   4. The donor disc is separated from the corneo-scleral donor tissue and placed endothelial side down or folded in half (if a 4.5mm incision was made) onto a healon coated transfer spatula.

      Transfer of donor to recipient

   1) Air is injected into the anterior chamber. 2) The donor tissue disc is placed into the anterior chamber through the lamellar incision.

   4) The spatula is removed from the eye by sliding out from under the Healon coating.

   5) The disc position is finely manipulated with a needle or hook as needed, taking care to minimize endothelial touch.

   5) The limbal wound is sutured with interrupted 10-0 nylon sutures. 6) The anterior chamber air bubble is replaced 50% with balanced salt solution. 7) A Seidel test is performed. If positive, additional limbal sutures are placed.

   8) The conjunctiva is closed with cautery or sutures. 9) Subconjunctival dexamethasone, 2 mg or Solu-Medrol, 30 mg and cefazolin, 25 mg or gentamicin, 20 mg, are injected in the inferior fornix. The eye is bandaged with a gauze patch and a Fox shield.

   10) The patient is instructed to spend the next two postoperative hours in a supine position.

   11) Routine postoperative orders for corneal transplantation are given upon discharge from the hospital that day.
   * PK The surgical method for patients randomized to penetrating keratoplasty will be the standard procedure currently practiced by the participating surgeons.

   POSTOPERATIVE CARE The patient will be seen the day after the surgery. Postoperative medications will include topical antibiotic of the surgeon?s choice, twice daily for one to two weeks and prednisolone acetate 1%, four times daily. The steroid drop will be tapered by one drop daily each month. Alterations to the steroid taper and other medical treatment will be made based upon individual patient conditions and response. Patient activity restrictions and eye protection measures will follow the usual PK recommendations by the individual surgeon. All patients will be seen at the following intervals: preoperatively and at 1 week (5-14 days), 1 month (3-6 weeks), 3 months (4-6 months), 6 months (5-7 months), and 1, 2, and 3 years (3 months) postoperatively. Keratograms will be performed at each visit, except one day and one week postoperatively. Confocal microscopy will be done as part of each keratogram and also at the one week postoperative visit. Additional clinic visits may be requested by the surgeon as needed for proper medical management. Corneal suture removal in penetrating grafts or limbal suture removal in DLEK will be dictated by patient healing and at the surgeon?s discretion.

   DATA COLLECTION AND STATISTICAL ANALYSIS Data collection will be performed with the instruments and schedule delineated above in the Methods section. The following outcome measures will be calculated from the data. These will be compared between the 2 groups (DLEK and PK) at each postoperative time by using t-tests or rank sum tests with Bonferroni corrections.

   Primary Outcome Measures
   1. Visual acuity with best refractive correction
   2. Refractive astigmatism
   3. Keratometric astigmatism
   4. Topographic astigmatism ("Simulated Keratometry" function of the TMS-1 mapping) Secondary Outcome Measures

   <!-- -->

   1. Corneal backscattered light
   2. Ocular forward-scattered light
   3. Contrast sensitivity
   4. Posterior corneal curvature
   5. Corneal sensitivity
   6. Corneal subbasal nerve density
   7. Keratocyte density
   8. Endothelial cell density
   9. Quality of visual function (NEI-VFQ) Statistical Power We have recently published variance data on keratometric astigmatism and endothelial cell density after PK. The keratometric astigmatism17 after removal of all sutures was 4.6  2.7 D (meanSD) and the endothelial cell density18 2 months postoperatively was 2606  446 cells/mm2. To detect (=0.05) a difference of 2.5 D in keratometric astigmatism with 80% certainty (=0.2) would require 20 subjects in each group, and to detect a difference of 400 cells/mm2 in endothelial cell density would require 20 subjects in each group. We expect to have 25 patients in each group, giving the study adequate power.

   For an additional use of the data, primary outcome data on the patients randomized to DLEK from our center will be pooled with data from other participating centers in the Endothelial Keratoplasty Group organized by Mark Terry, M.D., Portland, OR, who will coordinate data collection and statistical analysis. Pooled data will be used to calculate mean postoperative visual acuity, refractive outcomes and frequency of favorable outcome. These data will be compared with published data on PK.

ELIGIBILITY:
1. Corneal edema due to endothelial dysfunction
2. Aphakia, pseudophakia, or cataract requiring extraction
3. Visual acuity in a) study eye; best spectacle-corrected entrance acuity 20/40 or worse. b)contralateral eye; best spectacle-corrected entrance acuity equal to or better than the study eye and 20/200 or better.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Visual acuity.

SECONDARY OUTCOMES:
Astigmatism
contrast sensitivity
corneal haze
endothelial cell density
corneal thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Trousdale ER, Hodge DO, Baratz KH, Maguire LJ, Bourne WM, Patel SV. Vision-related quality of life before and after keratoplasty for Fuchs' endothelial dystrophy. Ophthalmology. 2014 Nov;121(11):2147-52. doi: 10.1016/j.ophtha.2014.04.046. Epub 2014 Jul 9. PMID 25015214
- [Derived] Ahuja Y, Baratz KH, McLaren JW, Bourne WM, Patel SV. Decreased corneal sensitivity and abnormal corneal nerves in Fuchs endothelial dystrophy. Cornea. 2012 Nov;31(11):1257-63. doi: 10.1097/ICO.0b013e31823f7888. PMID 22357383
- [Derived] McLaren JW, Patel SV, Bourne WM, Baratz KH. Corneal wavefront errors 24 months after deep lamellar endothelial keratoplasty and penetrating keratoplasty. Am J Ophthalmol. 2009 Jun;147(6):959-65, 965.e1-2. doi: 10.1016/j.ajo.2008.12.039. Epub 2009 Mar 19. PMID 19298950
- [Derived] Patel SV, McLaren JW, Hodge DO, Baratz KH. Scattered light and visual function in a randomized trial of deep lamellar endothelial keratoplasty and penetrating keratoplasty. Am J Ophthalmol. 2008 Jan;145(1):97-105. doi: 10.1016/j.ajo.2007.09.002. Epub 2007 Nov 8. PMID 17996211